CLINICAL TRIAL: NCT00850785
Title: A Pilot Study of Autologous Tumor DRibble Vaccine With Docetaxel in Stage IIIB and IV Non-Small Cell Lung Cancer
Brief Title: Autologous Tumor DRibble Vaccine in Patients With Non-Small Cell Lung Cancer
Acronym: DRibble
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: The Wayne D. Kuni and Joan E. Kuni Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-76; 1R21CA123864-01A2 (NIH)
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: DRibble vaccine — Docetaxel 75 mg/m2 will be administered in the several days after leukapheresis. Intradermal (ID) vaccine injections of DRibbles made from at least 5 million and up to 20 million cell equivalents per vaccination will begin 14 days after the first docetaxel. Each DRibble vaccine will be followed by the 6-day infusion of GM-CSF via the CADD-MS 3 pump (50 micrograms/24 hrs).

SUMMARY:
This is a pilot single institution study of DRibble vaccination + GM-CSF in patients with stage IIIB or IV NSCLC who have undergone 0-1 chemotherapy regimens for metastatic disease. The primary objective of this trial is to evaluate immune responses induced by autologous DRibble vaccine in vivo and in vitro and against autologous and allogeneic lung cancer cells.

DETAILED DESCRIPTION:
Ten patients will be enrolled. Study treatment is as follows: Docetaxel 75 mg/m2 will be given on day 1. Intradermal vaccinations of DRibbles from 5-20 x 106 cell equivalents per vaccine will begin 14 days after docetaxel. Immediately following vaccination, subcutaneous infusion of GM-CSF (50 micrograms/24 hrs) will be initiated. GM-CSF will be infused into the vaccination site for 6 days using the CADD-MS 3 pump.

A second docetaxel injection will be given at day 29 followed by a second vaccination 14 days later and 3 additional vaccines will be given at 2-week intervals. Following each vaccination, GM-CSF will again be infused over 6 days via the CADD-MS 3 pump.

Peripheral blood will be obtained for immune monitoring at each vaccination. DTH to autologous tumor and to DRibble vaccine will be tested before the first and fifth vaccines. A second leukapheresis for immune monitoring will be obtained at 12 weeks. Clinical tumor response will be assessed after the fifth vaccination unless clinical evidence of tumor progression occurs sooner.

Immune response will be assessed by DTH, T-cell function, T-cell migration into the vaccine sites and cytokine release assays. Sophisticated flow cytometry assays will be used to detect active T-cell subsets. Safety will be monitored by physical and laboratory exams at each vaccine visit and adverse events will be recorded and reported as appropriate. Clinical response will be assessed by tumor measurements by CT scan and/or physical exam at study entry and after 12 weeks. PFS and OS will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or IV NSCLC.
* Adequate pleural effusion (>600 cc) or subcutaneous metastases (>1 cc) for
* DRibble vaccine production.
* Measurable or evaluable disease.
* No or one prior chemotherapy regimen for advanced NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Age > 18 years.
* CD4 count > 200 per cc.
* Women of childbearing potential must have a negative pregnancy test and must avoid becoming pregnant while on treatment. Men must avoid fathering a child while on treatment. This exclusion is required due to the toxicities that docetaxel may have on the forming fetus, spermatogenesis or the nursing child.
* Also, because pregnancy may alter immune function it may limit the treatment efficacy.
* Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.

Anticipated lifespan minimum 6 months.

Exclusion Criteria:

* Prior vaccine or gene therapy for cancer.
* Untreated brain metastases or spinal cord compression.
* Active autoimmune disease.
* Active other malignancy.
* Known hypersensitivity to docetaxel.
* HIV positive and/or Hepatitis B or C positive.
* Patients receiving any other concurrent investigational treatment.
* Other medical or psychiatric conditions that in the opinion of the Principal
* Investigator would preclude safe participation in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Vaccine-induced immune response as measured by in vitro immune monitoring and by the delayed-type hypersensitivity (DTH) testing to injections of autologous, unmodified tumor cells and to DRibbles. | DTH on days 7-10 and days 77-80 and blood for immune monitoring (30-50 cc) prior to each vaccine.

SECONDARY OUTCOMES:
Tumor response (RECIST criteria) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Walter J Urba, MD, PhD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanborn RE, Ross HJ, Aung S, Acheson A, Moudgil T, Puri S, Hilton T, Fisher B, Coffey T, Paustian C, Neuberger M, Walker E, Hu HM, Urba WJ, Fox BA. A pilot study of an autologous tumor-derived autophagosome vaccine with docetaxel in patients with stage IV non-small cell lung cancer. J Immunother Cancer. 2017 Dec 19;5(1):103. doi: 10.1186/s40425-017-0306-6. PMID 29258618